CLINICAL TRIAL: NCT04141917
Title: Stepped-wedge Design Study of Point-of-care Molecular Testing for Influenza and Treatment With Baloxavir for Prevention of Secondary Transmission of Influenza in Homeless Shelters in Seattle, WA
Brief Title: Test-and-treat for Influenza in Homeless Shelters
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Operational futility (i.e. near zero circulation of influenza in the community during year 2)
Sponsor: University of Washington (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Helen Chu, Assistant Professor, School of Medicine: Division of Allergy & Infectious Diseases, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00007800
Record Dates: First submitted 2019-10-23; First posted 2019-10-28 (Actual); Results first posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-05

CONDITIONS: Influenza; Respiratory Viral Infection
Keywords: Tamiflu; Oseltamivir; Baloxavir; Influenza; Flu; Rapid Test; Xofluza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard influenza surveillance (No Intervention): Subjects exhibiting ≥ 2 ARI symptoms or new or worsening cough in the last 7 days at a participating shelter complete a survey collecting demographic and clinical data, and provide a mid-turbinate nasal swab for RT-PCR testing.
- Point-of-care molecular testing and treatment of influenza (Active Comparator): Subjects exhibiting ≥ 2 ARI symptoms, or new or worsening cough, in the last 48 hrs at a participating shelter complete a survey collecting demographic and clinical data, and provide a mid-turbinate nasal swab to be tested on-site with a molecular assay (Abbott ID NOW™ Influenza A & B (Chicago, IL)) and receive an antiviral if tested positive (XOFLUZA™ or Tamiflu®) .
  Interventions: Combination Product: Point-of-care molecular testing and treatment of influenza

INTERVENTIONS:
Combination Product: Point-of-care molecular testing and treatment of influenza — Eligible individuals will be tested on site with a point-of-care molecular influenza test and, if positive, offered antiviral treatment with baloxavir for those aged ≥12 years, or oseltamivir for those aged <12 years; pregnant; breastfeeding; liver disease; or are immunosuppressed. Follow-up nasal swabs and symptom diaries will be collected from participants 2 or 3 days after receiving the antiviral, and again 5, 6, or 7 days after receiving.
  Arms: Point-of-care molecular testing and treatment of influenza

SUMMARY:
This study is a stepped-wedge cluster-randomized trial of on-site rapid testing and treatment for influenza in homeless shelters within the Seattle area to determine whether this strategy reduced the incidence of influenza in the shelter environment.

DETAILED DESCRIPTION:
The study will be conducted over the course of two flu seasons, and all shelters will start with routine surveillance of influenza using mid-turbinate nasal swabs for sample collection and RT-PCR testing. Shelters will be randomized to implement a test-and-treat strategy at different months throughout flu season, treating individuals who present ARI symptoms or new or worsening cough within 2 days (48 hours). Shelters will continue routine surveillance until all offer the test-and-treat strategy. Eligible individuals will be tested on site with a point-of-care molecular influenza test and, if positive, offered antiviral treatment. Individuals with 3-7 days of symptoms, or who choose not to participate in the intervention strategy, will still be eligible for participation in the routine surveillance.

Our primary hypothesis is that implementation of a point-of-care diagnostic and antiviral treatment intervention among sheltered individuals experiencing homelessness will reduce the incidence of influenza within this population over the course of a flu season. A process evaluation will also be conducted to explore the feasibility of point-of-care testing implementation in this population.

ELIGIBILITY:
Inclusion Criteria:

* Resident for 1 or more days at a participating shelter
* ≥2 ARI symptoms or acute cough alone
* Willing to take study medication
* Willing to comply with all study procedures, including weekly surveillance and repeat nasal swab at day 2/3 and day 5/6/7 post-treatment
* Able to provide written, informed consent and/or assent

Exclusion Criteria:

* Any serious or uncontrolled medical disorder or active infection that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration
* Inability to consent and/or comply with study protocol
* Individuals who have received oseltamivir or baloxavir within past 7 days for treatment of influenza
* Individuals with known hypersensitivity to baloxavir marboxil or oseltamivir
* Individuals with chronic kidney disease

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1618 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Y Chu, MD, MPH, Principal Investigator — University of Washington
Locations (9):
- United States (9):
  - Mary's Place Burien, Burien, Washington
  - Compass Housing Alliance at First Presbyterian, Seattle, Washington
  - Downtown Emergency Service Center Shelter, Seattle, Washington
  - ROOTS Young Adult Shelter, Seattle, Washington
  - Compass Housing Alliance Blaine Center Men's Shelter, Seattle, Washington
  - Mary's Place North Seattle, Seattle, Washington
  - St Martin De Porres Shelter, Seattle, Washington
  - Compass Housing Alliance Jan & Peter's Place Women's Shelter, Seattle, Washington
  - Mary's Place White Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
We do not currently expect to share specimens with outside investigators, but if compelling opportunities arise that will advance the overall objectives of this research, the Executive Committee of the study will consider such requests. They alone have the authority to make such decisions.
  All biospecimens (nasal swabs) will be coded and identifiable through the study's main database. Any specimens shared with external investigators (if deemed appropriate by the Executive Committee) will have identifiers removed prior to sharing.

REFERENCES:
- [Background] Hayden FG, Sugaya N, Hirotsu N, Lee N, de Jong MD, Hurt AC, Ishida T, Sekino H, Yamada K, Portsmouth S, Kawaguchi K, Shishido T, Arai M, Tsuchiya K, Uehara T, Watanabe A; Baloxavir Marboxil Investigators Group. Baloxavir Marboxil for Uncomplicated Influenza in Adults and Adolescents. N Engl J Med. 2018 Sep 6;379(10):913-923. doi: 10.1056/NEJMoa1716197. PMID 30184455
- [Background] Boonyaratanakornkit J, Ekici S, Magaret A, Gustafson K, Scott E, Haglund M, Kuypers J, Pergamit R, Lynch J, Chu HY. Respiratory Syncytial Virus Infection in Homeless Populations, Washington, USA. Emerg Infect Dis. 2019 Jul;25(7):1408-1411. doi: 10.3201/eid2507.181261. PMID 31211675
- [Background] Hwang SW, Orav EJ, O'Connell JJ, Lebow JM, Brennan TA. Causes of death in homeless adults in Boston. Ann Intern Med. 1997 Apr 15;126(8):625-8. doi: 10.7326/0003-4819-126-8-199704150-00007. PMID 9103130
- [Background] Thiberville SD, Salez N, Benkouiten S, Badiaga S, Charrel R, Brouqui P. Respiratory viruses within homeless shelters in Marseille, France. BMC Res Notes. 2014 Feb 5;7:81. doi: 10.1186/1756-0500-7-81. PMID 24499605
- [Derived] Cox SN, Rogers JH, Thuo NB, Meehan A, Link AC, Lo NK, Manns BJ, Chow EJ, Al Achkar M, Hughes JP, Rolfes MA, Mosites E, Chu HY. Trends and factors associated with change in COVID-19 vaccination intent among residents and staff in six Seattle homeless shelters, March 2020 to August 2021. Vaccine X. 2022 Dec;12:100232. doi: 10.1016/j.jvacx.2022.100232. Epub 2022 Oct 19. PMID 36276877
- [Derived] Chow EJ, Casto AM, Roychoudhury P, Han PD, Xie H, Pfau B, Nguyen TV, Sereewit J, Rogers JH, Cox SN, Wolf CR, Rolfes MA, Mosites E, Uyeki TM, Greninger AL, Hughes JP, Shim MM, Sugg N, Duchin JS, Starita LM, Englund JA, Chu HY. The Clinical and Genomic Epidemiology of Rhinovirus in Homeless Shelters-King County, Washington. J Infect Dis. 2022 Oct 7;226(Suppl 3):S304-S314. doi: 10.1093/infdis/jiac239. PMID 35749582
- [Derived] Rogers JH, Cox SN, Hughes JP, Link AC, Chow EJ, Fosse I, Lukoff M, Shim MM, Uyeki TM, Ogokeh C, Jackson ML, Boeckh M, Englund JA, Mosites E, Rolfes MA, Chu HY. Trends in COVID-19 vaccination intent and factors associated with deliberation and reluctance among adult homeless shelter residents and staff, 1 November 2020 to 28 February 2021 - King County, Washington. Vaccine. 2022 Jan 3;40(1):122-132. doi: 10.1016/j.vaccine.2021.11.026. Epub 2021 Nov 15. PMID 34863618
- [Derived] Newman KL, Rogers JH, McCulloch D, Wilcox N, Englund JA, Boeckh M, Uyeki TM, Jackson ML, Starita L, Hughes JP, Chu HY; Seattle Flu Study Investigators. Point-of-care molecular testing and antiviral treatment of influenza in residents of homeless shelters in Seattle, WA: study protocol for a stepped-wedge cluster-randomized controlled trial. Trials. 2020 Nov 23;21(1):956. doi: 10.1186/s13063-020-04871-5. PMID 33228787
- [Derived] Rogers JH, Link AC, McCulloch D, Brandstetter E, Newman KL, Jackson ML, Hughes JP, Englund JA, Boeckh M, Sugg N, Ilcisin M, Sibley TR, Fay K, Lee J, Han P, Truong M, Richardson M, Nickerson DA, Starita LM, Bedford T, Chu HY; Seattle Flu Study Investigators. Characteristics of COVID-19 in Homeless Shelters : A Community-Based Surveillance Study. Ann Intern Med. 2021 Jan;174(1):42-49. doi: 10.7326/M20-3799. Epub 2020 Sep 15. PMID 32931328

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants for this test-and-treat intervention were recruited from homeless shelters across King County, WA and implemented over two respiratory virus seasons (11/15/2019 - 3/31/2020; 11/2/2020 - 3/31/2021). In Year 1, 9 shelters were randomized to receive the intervention in a stepped-wedge approach. Due to the impact of COVID-19, residents from 6 shelters were relocated to new facilities for social distancing reasons. Re-randomization, including these new facilities, occurred Year 2.
Pre-assignment Details: Since shelters were randomized to receive the intervention in cascading intervals as part of a stepped-wedge approach rather than participants themselves, participant study encounters rather than unique participants serve as the baseline unit of measure. Since participants are cross-sectionally recruited and not followed longitudinally unless they received antiviral treatment (for 1 week), there is no dropout between study periods, only new enrollments.
Units Other Than Participants: Shelters
Groups:
- Sequence A: 5 months of standard surveillance + test and treat protocol
  Standard influenza surveillance period: Subjects exhibiting ≥ 2 ARI symptoms or new or worsening cough in the last 7 days at a participating shelter complete a survey collecting demographic and clinical data, and provide a mid-turbinate nasal swab for RT-PCR testing.
  Point-of-care molecular testing and treatment of influenza period:
  Subjects exhibiting ≥ 2 ARI symptoms, or new or worsening cough, in the last 48 hrs at a participating shelter complete a survey collecting demographic and clinical data, and provide a mid-turbinate nasal swab to be tested on-site with a molecular assay (Abbott ID NOW™ Influenza A & B (Chicago, IL)) and receive an antiviral if tested positive (XOFLUZA™ or Tamiflu®) .
  Point-of-care molecular testing and treatment of influenza: Eligible individuals will be tested on site with a point-of-care molecular influenza test and, if positive, offered antiviral treatment with baloxavir for those aged ≥12 years, or oseltamivir for those aged <12 years; pregnant; breastfeeding; liver disease; or are immunosuppressed. Follow-up nasal swabs and symptom diaries will be collected from participants 2 or 3 days after receiving the antiviral, and again 5, 6, or 7 days after receiving.
- Sequence B: 1 month standard surveillance then 4 months standard surveillance + test and treat protocol
  Standard influenza surveillance period: Subjects exhibiting ≥ 2 ARI symptoms or new or worsening cough in the last 7 days at a participating shelter complete a survey collecting demographic and clinical data, and provide a mid-turbinate nasal swab for RT-PCR testing.
  Point-of-care molecular testing and treatment of influenza period:
  Subjects exhibiting ≥ 2 ARI symptoms, or new or worsening cough, in the last 48 hrs at a participating shelter complete a survey collecting demographic and clinical data, and provide a mid-turbinate nasal swab to be tested on-site with a molecular assay (Abbott ID NOW™ Influenza A & B (Chicago, IL)) and receive an antiviral if tested positive (XOFLUZA™ or Tamiflu®) .
  Point-of-care molecular testing and treatment of influenza: Eligible individuals will be tested on site with a point-of-care molecular influenza test and, if positive, offered antiviral treatment with baloxavir for those aged ≥12 years, or oseltamivir for those aged <12 years; pregnant; breastfeeding; liver disease; or are immunosuppressed. Follow-up nasal swabs and symptom diaries will be collected from participants 2 or 3 days after receiving the antiviral, and again 5, 6, or 7 days after receiving.
- Sequence C: 2 months standard surveillance then 3 months standard surveillance + test and treat protocol
  Standard influenza surveillance period: Subjects exhibiting ≥ 2 ARI symptoms or new or worsening cough in the last 7 days at a participating shelter complete a survey collecting demographic and clinical data, and provide a mid-turbinate nasal swab for RT-PCR testing.
  Point-of-care molecular testing and treatment of influenza period:
  Subjects exhibiting ≥ 2 ARI symptoms, or new or worsening cough, in the last 48 hrs at a participating shelter complete a survey collecting demographic and clinical data, and provide a mid-turbinate nasal swab to be tested on-site with a molecular assay (Abbott ID NOW™ Influenza A & B (Chicago, IL)) and receive an antiviral if tested positive (XOFLUZA™ or Tamiflu®) .
  Point-of-care molecular testing and treatment of influenza: Eligible individuals will be tested on site with a point-of-care molecular influenza test and, if positive, offered antiviral treatment with baloxavir for those aged ≥12 years, or oseltamivir for those aged <12 years; pregnant; breastfeeding; liver disease; or are immunosuppressed. Follow-up nasal swabs and symptom diaries will be collected from participants 2 or 3 days after receiving the antiviral, and again 5, 6, or 7 days after receiving.
- Sequence D: 3 months standard surveillance then 2 months standard surveillance + test and treat protocol
  Standard influenza surveillance period: Subjects exhibiting ≥ 2 ARI symptoms or new or worsening cough in the last 7 days at a participating shelter complete a survey collecting demographic and clinical data, and provide a mid-turbinate nasal swab for RT-PCR testing.
  Point-of-care molecular testing and treatment of influenza period:
  Subjects exhibiting ≥ 2 ARI symptoms, or new or worsening cough, in the last 48 hrs at a participating shelter complete a survey collecting demographic and clinical data, and provide a mid-turbinate nasal swab to be tested on-site with a molecular assay (Abbott ID NOW™ Influenza A & B (Chicago, IL)) and receive an antiviral if tested positive (XOFLUZA™ or Tamiflu®) .
  Point-of-care molecular testing and treatment of influenza: Eligible individuals will be tested on site with a point-of-care molecular influenza test and, if positive, offered antiviral treatment with baloxavir for those aged ≥12 years, or oseltamivir for those aged <12 years; pregnant; breastfeeding; liver disease; or are immunosuppressed. Follow-up nasal swabs and symptom diaries will be collected from participants 2 or 3 days after receiving the antiviral, and again 5, 6, or 7 days after receiving.
Period: Surveillance Year 1
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D
Started (This is all year 1 participants enrolled during standard surveillance months at their shelter of residence) | 63; 3 Shelters | 76; 2 Shelters | 81; 2 Shelters | 324; 2 Shelters
Completed | 63; 3 Shelters | 76; 2 Shelters | 81; 2 Shelters | 324; 2 Shelters
Not Completed | 0; 0 Shelters | 0; 0 Shelters | 0; 0 Shelters | 0; 0 Shelters
Period: Surveillance + Test and Treat Year 1
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D
Started (This is all year 1 participants enrolled during standard surveillance + test and treat protocol months at their shelter of residence) | 358; 3 Shelters | 153; 2 Shelters | 82; 2 Shelters | 83; 2 Shelters
Completed | 358; 3 Shelters | 153; 2 Shelters | 82; 2 Shelters | 83; 2 Shelters
Not Completed | 0; 0 Shelters | 0; 0 Shelters | 0; 0 Shelters | 0; 0 Shelters
Period: Summer Surveillance
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D
Started (This is all participants enrolled between 4/1/2020 and 11/1/2020 when only standard surveillance was conducted at all shelters as year 1 of the test and treat protocol took place between 11/15/2019 and 3/31/2020 and year 2 of the protocol took place between 11/2/2020 and 3/31/2021. Enrollments are noted as per their randomized shelter sequence from year 1.) | 73; 3 Shelters | 39; 2 Shelters | 54; 2 Shelters | 20; 2 Shelters
Completed | 73; 3 Shelters | 39; 2 Shelters | 54; 2 Shelters | 20; 2 Shelters
Not Completed | 0; 0 Shelters | 0; 0 Shelters | 0; 0 Shelters | 0; 0 Shelters
Period: Surveillance Year 2
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D
Started (This is all year 2 participants enrolled during standard surveillance months at their shelter of residence) | 3; 3 Shelters | 3; 2 Shelters | 10; 2 Shelters | 7; 2 Shelters
Completed | 3; 3 Shelters | 3; 2 Shelters | 10; 2 Shelters | 7; 2 Shelters
Not Completed | 0; 0 Shelters | 0; 0 Shelters | 0; 0 Shelters | 0; 0 Shelters
Period: Surveillance + Test and Treat Year 2
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D
Started (This is all year 1 participants enrolled during standard surveillance + test and treat protocol months at their shelter of residence) | 62; 3 Shelters | 13; 2 Shelters | 3; 2 Shelters | 3; 2 Shelters
Completed | 62; 3 Shelters | 13; 2 Shelters | 3; 2 Shelters | 3; 2 Shelters
Not Completed | 0; 0 Shelters | 0; 0 Shelters | 0; 0 Shelters | 0; 0 Shelters

BASELINE CHARACTERISTICS:
Groups:
- Standard Influenza Surveillance Period: Subjects exhibiting ≥ 2 ARI symptoms or new or worsening cough in the last 7 days at a participating shelter complete a survey collecting demographic and clinical data, and provide a mid-turbinate nasal swab for RT-PCR testing.
  These are all participants that enrolled when only standard surveillance, no intervention, was available at their shelter given the randomized sequence.
- Point-of-care Molecular Testing and Treatment of Influenza Period: Subjects exhibiting ≥ 2 ARI symptoms, or new or worsening cough, in the last 48 hrs at a participating shelter complete a survey collecting demographic and clinical data, and provide a mid-turbinate nasal swab to be tested on-site with a molecular assay (Abbott ID NOW™ Influenza A & B (Chicago, IL)) and receive an antiviral if tested positive (XOFLUZA™ or Tamiflu®) .
  Point-of-care molecular testing and treatment of influenza: Eligible individuals will be tested on site with a point-of-care molecular influenza test and, if positive, offered antiviral treatment with baloxavir for those aged ≥12 years, or oseltamivir for those aged <12 years; pregnant; breastfeeding; liver disease; or are immunosuppressed. Follow-up nasal swabs and symptom diaries will be collected from participants 2 or 3 days after receiving the antiviral, and again 5, 6, or 7 days after receiving.
  These are all participants that enrolled when both standard surveillance and the intervention was available at their shelter given the randomized sequence.
- Total: Total of all reporting groups
Arm/Group | Standard Influenza Surveillance Period | Point-of-care Molecular Testing and Treatment of Influenza Period | Total
Number analyzed (Participants) | 853 | 765 | 1618
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 85 | 62 | 147
  Between 18 and 65 years | 727 | 667 | 1394
  >=65 years | 41 | 36 | 77
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 521 | 576 | 1097
  Female | 323 | 181 | 504
  Other | 4 | 3 | 7
  Prefer not to say | 5 | 4 | 9
  Data missing | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 109 | 71 | 180
  Not Hispanic or Latino | 731 | 683 | 1414
  Unknown or Not Reported | 13 | 11 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 24 | 25 | 49
  Asian | 20 | 12 | 32
  Native Hawaiian or Other Pacific Islander | 14 | 2 | 16
  Black or African American | 231 | 191 | 422
  White | 370 | 355 | 725
  More than one race | 95 | 84 | 179
  Unknown or Not Reported | 99 | 96 | 195

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cases of Influenza in Shelters During the Intervention Period Compared to the Control Period
Description: The intervention period is when test and treatment on-site was available and the control period is when just standard surveillance was available at a shelter.
Time Frame: Year 1 of the intervention (4.5 months)
Population: Due to the impact of COVID-19 mitigation efforts on reduced influenza transmission in Year 2 of the study and subsequent early stop due to operational futility, the analysis population for the primary outcome only includes unique participants who enrolled in Year 1 of the study (11/15/19 - 3/31/20). For this primary outcome measure, we used the number of unique participants in Year 1 as the denominator rather than all participant enrollments.
Measure: Count of Participants; unit: Participants
Groups:
- Standard Influenza Surveillance Period: Subjects exhibiting ≥ 2 ARI symptoms or new or worsening cough in the last 7 days at a participating shelter complete a survey collecting demographic and clinical data, and provide a mid-turbinate nasal swab for RT-PCR testing.
- Point-of-care Molecular Testing and Treatment of Influenza Period: Subjects exhibiting ≥ 2 ARI symptoms, or new or worsening cough, in the last 48 hrs at a participating shelter complete a survey collecting demographic and clinical data, and provide a mid-turbinate nasal swab to be tested on-site with a molecular assay (Abbott ID NOW™ Influenza A & B (Chicago, IL)) and receive an antiviral if tested positive (XOFLUZA™ or Tamiflu®) .
  Point-of-care molecular testing and treatment of influenza: Eligible individuals will be tested on site with a point-of-care molecular influenza test and, if positive, offered antiviral treatment with baloxavir for those aged ≥12 years, or oseltamivir for those aged <12 years; pregnant; breastfeeding; liver disease; or are immunosuppressed. Follow-up nasal swabs and symptom diaries will be collected from participants 2 or 3 days after receiving the antiviral, and again 5, 6, or 7 days after receiving.
Arm/Group | Standard Influenza Surveillance Period | Point-of-care Molecular Testing and Treatment of Influenza Period
Number analyzed (Participants) | 363 | 371
Participants | 23 | 32
Statistical Analysis 1: Comparison: Standard Influenza Surveillance Period vs Point-of-care Molecular Testing and Treatment of Influenza Period; The number of influenza-positive tests was analyzed using a generalized linear mixed model following a Poisson distribution with a log link and robust variance. The model is adjusted for calendar time and an exposure time variable based on shelter capacity. This model includes symptomatic individuals who tested throughout Year 1 of the study (November 15, 2019 - March 31, 2020); Test type: Superiority; Risk Ratio, log = 1.33, 95% CI 2-sided [0.35 to 5.02]

2. Secondary Outcome: Feasibility of Implementation of Point-of-care Molecular Testing and Treatment of Influenza in Shelters
Description: Number of participants/participant encounters with les than 48 hours between symptom onset until diagnosis with RT-PCR.
Time Frame: Up to 24 months
Population: Includes all participant encounters from study Years 1 and 2. 153 participant encounters were missing this data because they were asymptomatic enrollments conducted once monthly at all shelters between 11/15/2019 and 3/31/2020.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Influenza Surveillance Period | Point-of-care Molecular Testing and Treatment of Influenza Period
Number analyzed (Participants) | 701 | 764
Participants | 266 | 308

3. Secondary Outcome: Feasibility of Implementation of Influenza Treatment in Shelters
Description: Number of influenza-positive participants identified through on-site molecular testing in the intervention period that were treated with an antiviral
Time Frame: Up to 24 months
Population: This outcome can only be assessed among participants enrollments from the intervention period as those in the control period ("standard influenza surveillance") were not eligible for antiviral treatment. Those that reported symptom onset ≥48 hours that were enrolled in the intervention period were dropped from the overall number of participants analyzed. The analysis population includes only influenza-positive cases that were detected using an on-site molecular test.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Influenza Surveillance Period | Point-of-care Molecular Testing and Treatment of Influenza Period
Number analyzed (Participants) | 0 | 21
Participants |  | 21

4. Secondary Outcome: Number of Participants That Drop Out of Study
Description: Measured as becoming lost to follow-up (did not complete both follow-up study visits on day 2/3 and day 5/6/7) after testing positive for influenza at baseline enrollment with an on-site molecular test and receiving an antiviral
Time Frame: Up to 24 months
Population: Only participant enrollments from the intervention period that tested positive for influenza at baseline enrollment with an on-site molecular test and received an antiviral are included in this analysis population as participant enrollments under the standard influenza surveillance period did not receive follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Influenza Surveillance Period | Point-of-care Molecular Testing and Treatment of Influenza Period
Number analyzed (Participants) | 0 | 21
Participants |  | 1

5. Secondary Outcome: Number of Participants That Show Non-compliance With Study Drug
Description: Only applicable to those that receive oseltamivir rather than baloxavir which is a single-dose antiviral. Measured based on self-report during follow-up visits with study research assistants. Non-compliance is measured as the participant self-reporting fewer doses taken than to be expected at time of of follow-up (e.g. a participant that took there first dose of oseltamivir in the AM on March 8 would be expected to have taken 6 doses if their follow-up visit was in the PM on March 10).
Time Frame: Up to 24 months
Population: This analysis population includes all participants that received oseltamivir as an antiviral and returned for at least one follow-up study visit when a number of doses of the medication was reported to study staff.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Influenza Surveillance Period | Point-of-care Molecular Testing and Treatment of Influenza Period
Number analyzed (Participants) | 0 | 6
Participants |  | 1

6. Secondary Outcome: Number of Laboratory-confirmed Influenza Cases That Report Fever
Description: Based on self-report of new or worsening fever in the past 7 days; not gold standard measurement
Time Frame: Up to 24 months
Population: All influenza positive cases detected in study Years 1 and 2; there were no cases of influenza detected in year 2 of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Influenza Surveillance Period | Point-of-care Molecular Testing and Treatment of Influenza Period
Number analyzed (Participants) | 23 | 32
Participants | 12 | 16

7. Secondary Outcome: Influenza Viral RNA Levels
Description: Measured mean cycle threshold (Ct) value for each laboratory-confirmed influenza-positive specimen collected at baseline enrollment, by subtype. Ct values have an inverse relationship with viral load.
Time Frame: Up to 24 months
Population: All influenza-positive specimen detected through RT-PCR in study Years 1 and 2. One individual in the standard surveillance period was coinfected with both Influenza A and Influenza B, therefore these row numbers are not mutually exclusive.
Measure: Mean (Inter-Quartile Range); unit: Cycle threshold value
Arm/Group | Standard Influenza Surveillance Period | Point-of-care Molecular Testing and Treatment of Influenza Period
Number analyzed (Participants) | 23 | 32
Cycle threshold value
  Influenza A: number analyzed (Participants) | 10 | 6
  Influenza A | 19.22 [16.50 to 22.19] | 21.21 [17.38 to 25.34]
  Influenza B: number analyzed (Participants) | 14 | 26
  Influenza B | 22.08 [18.47 to 26.26] | 18.51 [15.87 to 22.44]

8. Secondary Outcome: Number of Samples With Detectable Influenza RNA Virus at Days 2/3 and Days 5/6/7
Description: Measured at subject follow-up visits with nasal swabs provided to study staff; provided subject has not become lost to follow up.
Time Frame: Up to 24 months
Population: Only includes influenza-positive samples from participant enrollments collected in the intervention period and detected with an on-site molecular test. Of the 21 participants that received an antiviral and, according to the protocol, should have returned for follow-up sample collect and study visits, only 14 returned on day 2/3 and only 1 returned for day 2/3 and day 5/6/7 study visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Influenza Surveillance Period | Point-of-care Molecular Testing and Treatment of Influenza Period
Number analyzed (Participants) | 0 | 21
Participants
  Detectable at day 2/3: number analyzed (Participants) | 0 | 14
  Detectable at day 2/3 |  | 7
  Detectable at day 5/6/7: number analyzed (Participants) | 0 | 1
  Detectable at day 5/6/7 |  | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the intervention periods implemented over two respiratory virus seasons: 11/15/19 - 3/31/20 and 11/2/20 - 3/31/21 (9 months total)
Description: Adverse event data, including symptom logs, were collected from trial participants that had follow-up visits 2/3 days and 5/6/7 days post-treatment. Adverse event data was not systematically collected from standard surveillance participants or from participants in the intervention period that did not participate in the trial component (on-site testing plus receipt of antiviral of influenza-positive).
Arm/Group | Standard Influenza Surveillance Period | Point-of-care Molecular Testing and Treatment of Influenza Period
All-Cause Mortality (participants affected / at risk) | 0/853 | 0/765
Serious Adverse Events (participants affected / at risk) | 0/853 | 0/765
Other Adverse Events (participants affected / at risk) | 0/853 | 5/765
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Influenza Surveillance Period (N=853) | Point-of-care Molecular Testing and Treatment of Influenza Period (N=765)
Nausea or vomiting (Gastrointestinal disorders) | 0 | 2
Ear pain or ear discharge (Ear and labyrinth disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasopharyngitis (General disorders) | 0 | 1
Headache (General disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Inflamed mucous membrane (Immune system disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Decline in influenza activity following the advent of SARS-CoV-2 public health mitigation measures led to early termination of study for operational futility purposes. Low infection detection and study power after year 1 also limited our ability to conduct statistical analyses on several intended secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT04141917/Prot_SAP_000.pdf